CLINICAL TRIAL: NCT06908512
Title: Turkish Adaptation, Validity and Reliability of the Intensive Care Unit-specific Pressure Injury Risk Assessment Scale
Brief Title: Adaptation of the Intensive Care Unit-specific Pressure Injury Risk Scale to Turkish (RAPS-ICU)
Status: Not yet recruiting | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, İbrahim Caner Di̇ki̇ci̇, Assist. Prof., Harran University
Other Study IDs: NT268347145
Record Dates: First submitted 2025-03-19; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Pressure Injury; Reliability and Validity; Intensive Care Units (ICUs); Assessment Scale
Keywords: Pressure Injury; Reliability and Validity; Intensive Care Units; Assessment Scale
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study was to evaluate the translation, cross-cultural fit, and psychometric properties of the ICU-specific pressure injury risk scale

DETAILED DESCRIPTION:
This was a prospective, cross-sectional study aimed at translation and cultural adaptation of the RAPS-ICU into Turkish, while also assessing its validity and reliability.Patients who meet the inclusion criteria and who are hospitalized in the Intensive Care Clinics of Istinye University Bahçeşehir Liv Hospital and Harran University Hospital will participate in the study. In this study, Turkish adaptation of the 'Intensive care unit-specific pressure injury risk assessment scale' is planned. After language adaptation, its validity and reliability will be tested. The reliability of the intensive care unit-specific pressure injury risk assessment scale will be assessed by inter-rater reliability and internal consistency (determined by calculating Cronbach alpha coefficient), and its validity will be assessed by convergent and divergent validity of the scale. Relative reliability was obtained by calculating the intraclass correlation coefficient (ICC). Relative reliability will be obtained by calculating the intraclass correlation coefficient (ICC). The receiver operator characteristics (ROC) curve has been used to estimate sensitivity and specificity and will represent the false positive rate versus the true positive rate across various thresholds for different scores.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Staying in the Intensive Care Unit for at least 1 day,
* Agreeing to participate in the study by themselves or a family member.
* Volunteering to participate in the research
* Full orientation and no psychiatric problems

Exclusion Criteria:

- Having communication problems

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients in intensive care units
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2025-07-12 (Estimated); Study Completion 2025-11-12 (Estimated)

PRIMARY OUTCOMES:
ICU-Specific Pressure Injury Risk Assessment Scale (RAPS-ICU) | Baseline
  The RAPS-ICU was developed by W°ahlin et al to identify patients at risk of developing pressure injuries in the ICU. The RAPS-ICU has six domains that assess failure in vital organs, mobility, moisture, sensory perceptions, special treatments, and consciousness. Five of the six domains scored 1-4 points progressing from most to least severity of alteration; failure in vital organs domains ranged from 1-3 points. Overall PI risk is reflected by a total score ranging from 6 to 23. The lower the total score the greater the estimated risk of developing a PI. Risk scores can be categorized as increased (16-18), high (12-15), and very high (≤11) risk for PI.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Şahin, Assist. Prof., Study Chair — Harran University
Locations (1):
- Harran University, Sanliurfa, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wahlin I, Ek AC, Lindgren M, Geijer S, Arestedt K. Development and validation of an ICU-specific pressure injury risk assessment scale. Scand J Caring Sci. 2021 Sep;35(3):769-778. doi: 10.1111/scs.12891. Epub 2020 Jul 14. PMID 32666602